CLINICAL TRIAL: NCT01357083
Title: The Study of Morning and Nocturnal Serum Melatonin Rhythm Levels in Patients With Major Depressive Disorder
Brief Title: The Study of Serum Melatonin Rhythm Levels in Patients With Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: Science & Research Islamic Azad University Branch Khozestan (Other)
Responsible Party: shahnaz Khaleghipour, Science & Research Islamic Azad University Branch Khozestan
Other Study IDs: 9460; CCT-NAPN-21087
Record Dates: First submitted 2011-05-10; First posted 2011-05-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2009-08

CONDITIONS: Major Depressive Disorder
Keywords: Melatonin; Periodicity; Depressive disorder, major; Serum; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Major Depression Disorder: This study is analytical cross-sectional and randomized. Two groups of depressed patients and healthy subjects were selected.The individual were submitted to a medical examination, and responded to the Beck depression inventory (BDII-II). Those, who got a score above 20, were included in the depressed group. Among this group, 50 patients were chosen randomly. those who obtained a depressive score below 9, 50 of them were chosen and they were included in the healthy group. The control group was chosen to match to the depressed patients for education, social occasion, occupational and economical situation. All of the subjects were interviewed psychiatrically, and the depression disorder was confirmed on the basis of the DSM criteria. eight out of 50 depressed patients were excluded from the study due to suffering from other psychiatric disorders .

SUMMARY:
One of the main points in the biological trends is, the circadian rhythm and disturbance in this cycle, which cause mood disorders and irregularity in this bio clock, to get depression. The pineal gland with the precise regulation of circadian rhythm of melatonin regulates the brain haemostasis. The abnormal function of this gland gives rise to psychiatric disorders.

In the period of youth and early of middle-age cause biochemical changes and disturbance in biorhythm including melatonin secretion.

This process can change the peak of melatonin phase. In addition, a decrease in the level of serum melatonin, can change the function of immune system of depressed patients. This function facilitates the process of cancerous cell formation and tumor growth.

With respect to the conflicting results and that the positive and negative roles of melatonin in the creation of depression is unknown, the aim of this study was to compare the morning and nocturnal serum melatonin rhythm levels in the patients with Major Depressive Disorder. The second purpose was to measure the morning and nocturnal serum melatonin levels in the depressed and healthy men and women.

ELIGIBILITY:
Inclusion Criteria:

1. age: 22-48 years old
2. gender: male, female
3. who got a depressive score above 20, were included in the depressed group
4. those who obtained a depressive score below 9, were chosen and they were included in the healthy control group.
5. the healthy control group to match to the depressed patients for education, social occasion, occupational and economical situation.
6. the depression disorder was confirmed on the basis of the DSM criteria

Exclusion Criteria:

1. present or past psychiatric
2. physical diagnoses
3. drug consumption
4. use of narcotic substances
5. physical and psychosomatic disorders
6. the stressor
7. malfunction of thyroid gland
8. shift working

Ages: 22 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The individuals were chosen who referred to the industrial medical unit of one of big company.
Sampling Method: Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Depression status(measured by Beck depression inventory (BDII-II)) | 2weeks

SECONDARY OUTCOMES:
Measurements of morning and nocturnal melatonin levels by ELISA kit (cat no. RE54021) from the IBL-Hamburg. | 1 week
  The blood vein (5 milliliters) was taken from two groups at 8:00 am on a particular day. At the end of the same day and 24:00 h, the subjects were retaken the blood samples under the dim light.

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz Khaleghipour, PhD, Principal Investigator — Science and Research Branch Islamic Azad University Khozestan
Locations (1):
- Shahnaz Khaleghipour, Isfahan, Isfahan, Iran

REFERENCES:
- [Derived] Khaleghipour S, Masjedi M, Ahade H, Enayate M, Pasha G, Nadery F, Ahmadzade G. Morning and nocturnal serum melatonin rhythm levels in patients with major depressive disorder: an analytical cross-sectional study. Sao Paulo Med J. 2012;130(3):167-72. doi: 10.1590/s1516-31802012000300006. PMID 22790549